CLINICAL TRIAL: NCT01841658
Title: Effect of Obesity and Folic Acid Supplementation on Gene-specific DNA Methylation in Women of Reproductive Age
Brief Title: Folic Acid Supplementation in Women of Child Bearing Age
Acronym: FASUPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Georgia (Other)
Collaborators: University of Florida (Other); Emory University (Other)
Responsible Party: Principal Investigator, Lynn B. Bailey, PhD, Department Head and Professor, University of Georgia
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: UGA_FASUPPLEMENT_EPIGEN
Record Dates: First submitted 2013-04-19; First posted 2013-04-26 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-07

CONDITIONS: Obesity
Keywords: Folate Status; Folate Biomarkers
MeSH Terms: conditions — Obesity | interventions — Folic Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Folic Acid Normal Weight (Experimental): Folic acid, tablet, 800 mcg, daily, eight weeks. Normal Weight individuals, each will serve as her own control.
  Interventions: Dietary Supplement: Folic acid
- Folic acid Obese (Experimental): Folic acid, tablet, 800 mcg, daily, eight weeks. Obese individuals, each will serve as her own control.
  Interventions: Dietary Supplement: Folic acid

INTERVENTIONS:
Dietary Supplement: Folic acid — Participants will be instructed to consume 2 tablets per day, a total of 800 micrograms folic acid. To facilitate compliance, participants will be instructed in the use of a compliance calendar and will receive frequent telephone and 'text' reminders from project staff. Additionally, compliance will be determined by return pill count.

SUMMARY:
The objective of this study is to identify genes whose expression is potentially modifiable due to changes in folate intake and help delineate mechanisms accounting for the variability in individual response to folic acid supplementation. The study will be conducted in normal weight and obese women of childbearing age, supplemented for 8 weeks with 800 mcg/day folic acid.

It is hypothesized that (1) a change in folate status, induced by the supplementation, will influence the DNA methylation of specific genes and (2) the DNA methylation response to folic acid supplementation may differ between the normal weight and the obese women of childbearing age.

DETAILED DESCRIPTION:
This study will be conducted in two phases. An initial screening study will be performed to determine folate status, MTHFR677 genotype and body composition of potential participants of the intervention study. Both folate status and MTHFR677 genotype are known independent predictors of response to folic acid supplementation. Blood samples will be collected, after an overnight fast, for determination of serum folate concentration and for MTHFR677 genotyping. Body composition and 24-hr dietary recalls will also be conducted during the screening visit.

The second phase is an eight week supplementation trial with 800 mcg/day folic acid. Screened individuals determined to have a serum folate < 30 nmol/L (< 50th percentile of NHANES 1999-2004) and of the CC or CT genotype (for MTHFR677) will be eligible for inclusion in the supplementation trial. Participants will be instructed to avoid dietary supplements, fortified ready-to-eat cereals, and other high folate content foods during intervention. Blood samples will be collected, after an overnight fast, at baseline and after 4 and 8 weeks of supplementation for determination of primary (DNA methylation profile) and secondary (nutritional, metabolic and health status biomarkers) outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Screening Phase:
* Female 18-40 yr
* Body Mass index 18.5 to 24.9 or > 30 kg/m2
* Intervention Study:
* Serum folate < 30 nmol/L
* MTHFR677CC or MTHFR677CT genotype

Exclusion Criteria:

* Currently pregnant, pregnancy within past 12 months
* Greater than 2 previous pregnancies
* Use of prescription drugs other than oral contraceptives
* Chronic disease (diabetes, hypertension,epilepsy,cancer, kidney disease, CVD)
* Acute illness (pneumonia, urinary tract infection, mononucleosis)
* Use of antibiotics in past 30 days
* Current smoker
* Use of dietary supplements including multivitamins in past 30 days
* Habitual consumption of fortified ready-to-eat cereals
* Significant weight change in past 12 months
* Typical alcohol consumption of 2 or more drinks per day
* INTERVENTION: all above plus serum folate > 30 nmol/L; MTHFR677TT genotype

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2013-04; Primary Completion 2015-08 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Cell-type-specific DNA methylation | Baseline, 4 weeks and 8 weeks
  Change in DNA methylation in response to 4 or 8 weeks supplementation with 800 mcg/day of folic acid will be determined in DNA isolated from specific white blood cell types. Microarray analysis will be used to assess changes in multiple methylation sites within regulatory pathways for folate metabolism and/or development. Each subject will serve as her own control.
Gene-specific DNA methylation | Baseline, 4 weeks and 8 weeks
  Change in DNA methylation in response to 4 or 8 weeks supplementation with 800 mcg/day of folic acid will be determined in DNA isolated from whole blood . Microarray analysis will be used to assess changes in multiple methylation sites of specific genes within regulatory pathways for folate metabolism and/or development. Each subject will serve as her own control.

SECONDARY OUTCOMES:
Serum folate | Baseline, 4 weeks and 8 weeks
  Change in serum folate concentrations in response to 4 or 8 weeks supplementation with 800 mcg/day of folic acid will be determined by microbiological assay using Lactobacillus rhamnosus. Each subject will serve as her own control.
Red Blood Cell (RBC) Folate | Baseline, 4 weeks and 8 weeks
  Change in red blood cell (RBC) folate in response to 4 or 8 weeks supplementation with 800 mcg/day of folic acid will be determined by microbiological assay using Lactobacillus rhamnosus.
Body Composition | Baseline and 8 weeks
  Body composition in terms of fat mass (g), lean mass (g) and % body fat will be determined using the BODPOD instrument and verified by dual-energy X-ray absorptiometry (DXA). The DXA analysis will also provide an indication of regional fat distribution, and total bone area, bone mineral content and bone density.

CONTACTS AND LOCATIONS:
Overall Officials: Lynn B Bailey, PhD, Principal Investigator — University of Georgia; Dorothy Hausman, PhD, Study Director — University of Georgia
Locations (1):
- University of Georgia, Athens, Georgia, United States